CLINICAL TRIAL: NCT00005163
Title: Validation and Field Test for Risk Appraisal Instruments
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1035; R01HL032141 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Heart Disease Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To field test the validity, reliability, cost, and cost-benefit of Health Risk Appraisal (HRA) instruments.

DETAILED DESCRIPTION:
BACKGROUND:

Health Risk Appraisals instruments have provided the field of health promotion with an imaginative motivational and instructional tool to foster personal behavioral change. A HRA typically asked questions about smoking, blood pressure, exercise, medical history, diet and other life style variables. These risk indicators were then compared to epidemiological and mortality data to yield an estimate of an individual or group's risk for disease. They were widely regarded as the most promising new addition to the health promotion armamentarium. The National Health Information Clearinghouse divided them into the following three categories: Computer-Scored HRAs, which were mailed to a central computer facility for batch processing and were usually the more complex and detailed appraisals; Microcomputer-Based HRAs, which c;ould be processed by a microcomputer at home, in schools or at the worksite; and Self-Scored HRAs, which were usually brief, did not involve a computer, and were scored by the user.

Although HRAs were a burgeoning industry in health education, no properly designed and conducted scientific evaluation of them on a sufficiently large and representative sample of the general population had been undertaken in the United States or elsewhere.

DESIGN NARRATIVE:

In the first stage, fourteen HRAs were evaluated by determining the validity of the scoring system for estimating cardiovascular risk as employed in the Framingham Heart Study data base, the accuracy of the reported risk factor scores as measured by physiological values, and the understandability and social acceptability of the instrument format. The second stage of the project was a field test to determine reliability and cost-effectiveness. Ten groups of respondents were formed by randomly assigning eligible adults to one of the five HRA groups and then to reliability and validity status.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1983-09; Study Completion 1989-05 (Actual)

REFERENCES:
- [Background] Washburn RA, Goldfield SR, Smith KW, McKinlay JB. The validity of self-reported exercise-induced sweating as a measure of physical activity. Am J Epidemiol. 1990 Jul;132(1):107-13. doi: 10.1093/oxfordjournals.aje.a115622. PMID 2192545
- [Background] Avis NE, McKinlay JB, Smith KW. Is cardiovascular risk factor knowledge sufficient to influence behavior? Am J Prev Med. 1990 May-Jun;6(3):137-44. PMID 2397137
- [Background] Smith KW, McKinlay SM, Thorington BD. The validity of health risk appraisal instruments for assessing coronary heart disease risk. Am J Public Health. 1987 Apr;77(4):419-24. doi: 10.2105/ajph.77.4.419. PMID 3826459
- [Background] Smith KW, McKinlay SM, McKinlay JB. The reliability of health risk appraisals: a field trial of four instruments. Am J Public Health. 1989 Dec;79(12):1603-7. doi: 10.2105/ajph.79.12.1603. PMID 2817186
- [Background] Avis NE, Smith KW, McKinlay JB. Accuracy of perceptions of heart attack risk: what influences perceptions and can they be changed? Am J Public Health. 1989 Dec;79(12):1608-12. doi: 10.2105/ajph.79.12.1608. PMID 2817187